CLINICAL TRIAL: NCT01971476
Title: Open, Non-controlled, Dose Escalating Phase I Trial to Evaluate the Pharmacokinetics, Pharmacodynamics, Tolerability and Toxicity of Volasertib in Paediatric Patients From 2 Years to Less Than 18 Years of Age With Acute Leukaemia or Advanced Solid Tumour, for Whom no Effective Treatment is Known
Brief Title: Open Dose Escalating Trial to Determine the Maximum Tolerated Dose in Paediatric Patients With Advanced Cancers for Whom no Therapy is Known
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.27; 2013-001291-38 (EudraCT Number)
Record Dates: First submitted 2013-10-10; First posted 2013-10-29 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Leukemia; Neoplasms
MeSH Terms: conditions — Leukemia; Neoplasms | interventions — BI 6727

ARMS (1):
- All patients (Experimental): Volasertib will be administered as intravenous infusion
  Interventions: Drug: volasertib

INTERVENTIONS:
Drug: volasertib — intravenous administration on day 1of a treatment course

SUMMARY:
The present trial will be performed according to an open design to determine the maximum tolerable dose (MTD) by evaluation of dose-limiting toxicity (DLT) of volasertib in paediatric leukaemia and solid tumours in the age group 2 to less than 12 and 12 to less than 18 years. A further objective is to collect data on safety, tolerability, toxicity, efficacy (preliminary activity), pharmacokinetics and pharmacodynamics of volasertib in paediatric cancer patients

ELIGIBILITY:
Inclusion criteria:

* paediatric patients with leukaemia or advanced solid tumours including lymphomas (age 2 - less than 18 years) for whom no further treatment is known
* Lansky score > 60 for children 2 to less than 12 years
* Karnofsky score > 60 for children aged 12 or older
* life expectancy of at least 6 weeks as judged by the investigator
* parents or legal guardians have given written informed consent and informed assent suitable for the respective age group obtained

Exclusion criteria:

* patient eligible for other anti-leukaemic therapy with curative intent or effective therapy known for solid tumour therapy
* presence of cardiac disease (LVEF by echocardiography less than 25 %)
* symptomatic Central Nervous System involvement of the malignant disease
* primary CNS tumour
* inadequate lab parameters
* inadequate venous access
* QTc prolongation
* pregnancy, breastfeeding
* other diseases or CTs that might interfere with evaluation of safety

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- UNIV UZ Gent, Ghent, Belgium
- University Hospital Motol, Prague, Czechia
- INS Curie, Paris, France
- Universitätsklinikum Köln (AöR), Cologne, Germany
- Osp. Pediatrico Bambin Gesù, Roma, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the age group 2 to <12 years, 12 patients were entered and treated. In the age group 12 to <18 years, 10 patients were entered and treated.
Pre-assignment Details: In the age group 2 to <12 years, 15 patients were screened, with 3 screen failures. In the age group 12 to <18 years, 14 patients were screened, with 4 screen failures.
Groups:
- Volasertib 200 mg/m2: The patients were administered Volasertib 200 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour (h) on Day 1 of 14-day cycle.
- Volasertib 250 mg/m2: The patients were administered Volasertib 250 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour on Day 1 of 14-day cycle.
- Volasertib 300 mg/m2: The patients were administered Volasertib 300 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour on Day 1 of 14-day cycle.
Period: Cohort 1: 2 to <12 Years
Arm/Group | Volasertib 200 mg/m2 | Volasertib 250 mg/m2 | Volasertib 300 mg/m2
Started | 3 | 3 | 6
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 6
Not completed — Other not defined | 3 | 3 | 6
Period: Cohort 2: 12 to <18 Years
Arm/Group | Volasertib 200 mg/m2 | Volasertib 250 mg/m2 | Volasertib 300 mg/m2
Started | 6 | 4 | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 4 | 0
Not completed — Other not defined | 6 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: The treated set consisted of all patients who have received at least 1 dose of trial medication at the time of clinical cut-off.
  2 to <12 years (N=3, 3, 6). 12 to < 18 years (N=6, 4, 0).
Groups:
- Volasertib 200 mg/m2: The patients were administered Volasertib 200 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour on Day 1 of 14-day cycle.
- Total: Total of all reporting groups
Arm/Group | Volasertib 200 mg/m2 | Volasertib 250 mg/m2 | Volasertib 300 mg/m2 | Total
Number analyzed (Participants) | 9 | 7 | 6 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years]
  2 to <12 years | 7.0 (3.6) | 6.3 (3.1) | 7.0 (3.3) | 6.8 (3.0)
  12 to <18 years | 14.3 (2.3) | 15.8 (1.5) | NA (NA) — No patients entered. | 14.9 (2.1)
Sex/Gender, Customized [Number; unit: Participants]
  Female (2 to <12 years) | 1 | 2 | 3 | 6
  Male (2 to <12 years) | 2 | 1 | 3 | 6
  Female (12 to <18 years) | 2 | 0 | 0 | 2
  Male (12 to <18 years) | 4 | 4 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in the First Cycle for the Determination of the Maximum Tolerated Dose (MTD)
Description: This outcome measure presents number of participants with DLTs in the first cycle for the determination of MTD. DLTs were defined as drug related Common Terminology Criteria for Adverse Events (CTCAE) ≥Grade 3 (haematological and nonhaematological) Adverse Events (AEs) with the exception of a) Reduced blood cell count (any grade) without associated clinical complications qualifying for DLT. b) Febrile neutropenia Grade 3. c) Infection Grade 3 with neutrophil count <1000/mm3. d) Uric acid Grade ≥3. e) Nausea, vomiting and/or diarrhoea managed by adequate therapy (i.e. recovery to CTCAE Grade ≤2).
Time Frame: Up to 14 days.
Population: Treated Set: The treated set consisted of all patients who have received at least 1 dose of trial medication at the time of clinical cut-off.
Measure: Number; unit: Participants
Groups:
- 2 to <12 Years: Volasertib 200 mg/m2; 12 to <18 Years: Volasertib 200 mg/m2: The patients were administered Volasertib 200 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour on Day 1 of 14-day cycle.
- 2 to <12 Years: Volasertib 250 mg/m2; 12 to <18 Years: Volasertib 250 mg/m2: The patients were administered Volasertib 250 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour on Day 1 of 14-day cycle.
- 2 to <12 Years: Volasertib 300 mg/m2; 12 to <18 Years: Volasertib 300 mg/m2: The patients were administered Volasertib 300 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour on Day 1 of 14-day cycle.
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 4 | 0
Participants | 0 | 0 | 0 | 0 | 2 |

2. Primary Outcome: Maximum Tolerated Dose of Volasertib
Description: This outcome measure presents MTD of Volasertib. The MTD was defined as the highest dose level at which DLTs were reported in not more than 1 in 6 evaluable patients during Cycle 1.
Time Frame: Up to 14 days.
Population: as for outcome 1
Measure: Number; unit: mg
Arm/Group | 12 to <18 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2
Number analyzed (Participants) | 12 | 10
mg | 300 | 200

3. Secondary Outcome: Number of Patients With Hepatic Injury Defined as Adverse Events of Special Interest (AESI)
Description: This outcome measure presents number of patients with hepatic injury defined as AESI. Hepatic injury was defined by the following alterations of liver parameters: an elevation of Aspartate Transaminase (AST) and/or Alanine Transaminase (ALT) >3x Upper Limit of Normal (ULN) combined with an elevation of total bilirubin >2x ULN measured in the same blood sample.
Time Frame: Up to 879 days.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 4 | 0
Participants
  Total AEs in grouped category hepatic impairment | 0 | 1 | 1 | 3 | 1 |
  Alanine aminotransferase increased | 0 | 1 | 0 | 2 | 0 |
  Aspartate aminotransferase increased | 0 | 1 | 0 | 0 | 0 |
  Blood alkaline phosphatase increased | 0 | 0 | 1 | 0 | 0 |
  Metabolism and nutrition disorders | 0 | 0 | 0 | 0 | 1 |
  Hypoalbuminaemia | 0 | 0 | 0 | 0 | 1 |
  Hepatobiliary disorders | 0 | 0 | 0 | 1 | 0 |
  Hyperbilirubinaemia | 0 | 0 | 0 | 1 | 0 |
  Blood bilirubin increased | 0 | 0 | 0 | 1 | 0 |
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 1 | 0 |

4. Secondary Outcome: Number of Patients With Clinically Relevant Laboratory Value Changes of Calcium (Hyper- and/or Hypocalcaemia) as Judged by the Investigator and Reported as AEs, CTCAE Grade ≥3
Description: This outcome measure presents number of patients with clinically relevant laboratory value changes of calcium (hyper- and/or hypocalcaemia) as judged by the investigator and reported as AEs, CTCAE Grade ≥3. CTCAE Grade 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: Up to 879 days.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 4 | 0
Participants
  Total AEs clinically relevant changes of calcium | 0 | 0 | 0 | 0 | 0 |
  Metabolism and nutrition disorders | 0 | 0 | 0 | 0 | 0 |
  Hypocalcaemia | 0 | 0 | 0 | 0 | 0 |
  Hypercalcaemia | 0 | 0 | 0 | 0 | 0 |

5. Secondary Outcome: The Number of Patients With Changes in Cardiac Activity (Prolonged QTc Interval) Reported as Clinically Relevant Observations
Description: This outcome measure presents the number of patients with changes in cardiac activity (prolonged QTc interval) reported as clinically relevant observations to assess cardiac activity based on Electrocardiogram (ECG) recordings (digital, triplicate) before and at the end of each Volasertib administration and at least at 2 more time points within the first 24 hours after end of the first Volasertib administration. Two methods of heart rate correction of the QT interval were used: the fixed corrections Fridericia's correction (QTcF) and Bazett's correction (QTcB).
  SMQ: Standardised Medical Dictionary for Regulatory Activities (MedDRA) query.
Time Frame: Up to 879 days.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 4 | 0
Participants
  Total AEs in the MedDRA SMQ of QT prolongation | 0 | 0 | 1 | 2 | 1 |
  Electrocardiogram QT prolonged | 0 | 0 | 1 | 1 | 1 |
  Cardiac disorders | 0 | 0 | 0 | 1 | 0 |
  Conduction disorder | 0 | 0 | 0 | 1 | 0 |

6. Secondary Outcome: Best Overall Response [in Leukaemia Patients]: (Complete Remission (CR)), CR With Incomplete Neutrophil or Platelet Recovery (CRi), Partial Remission (PR), Stable Disease (SD), Progressive Disease (PD) and Death in Aplasia
Description: This outcome measure includes, CR: Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary (EM) disease; absolute neutrophil count ≥ 1.0 x 109/L (1000/μL); platelet count ≥80 x 109/L (80000/μL); independence of red blood cells transfusions. CRi: All CR criteria except for residual neutropenia (<1.0 x 109/L [1000/μL]) or thrombocytopenia (<800 x 109/L [80000/μL]), independence of red blood cell transfusions not required. PR: Decrease of bone marrow blast percentage to 5%-25%; decrease of pretreatment bone marrow (baseline) blast percentage by at least 50%; absence of EM disease. SD: Neither qualifies for CR, CRi, PR or PD. PD: At least one of the criteria a) 50% increase in bone marrow blast count over baseline b) 50% increase in peripheral blast count over baseline - evidence of new EM disease - clinically PD based on the judgment of the investigator. Death in aplasia: Deaths occurring ≥7 days after last administration of the trial drug while cytopenic.
Time Frame: Up to 849 days.
Population: Treated Set: The treated set consisted of all patients who have received at least 1 dose of trial medication at the time of clinical cut-off.
  The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Measure: Number; unit: Participants
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 2 | 2 | 0 | 2 | 1 | 0
Participants
  Complete remission | 0 | 0 |  | 0 | 0 |
  CRi* | 0 | 0 |  | 0 | 0 |
  Partial remission | 0 | 0 |  | 0 | 0 |
  Stable disease | 2 | 2 |  | 1 | 0 |
  Progressive disease | 0 | 0 |  | 1 | 1 |
  Death in aplasia | 0 | 0 |  | 0 | 0 |
  Not evaluable | 0 | 0 |  | 0 | 0 |
  Missing | 0 | 0 |  | 0 | 0 |

7. Secondary Outcome: Event-Free Survival (EFS) [in Leukaemia Patients]
Description: EFS was defined as the time from the first infusion of Volasertib to the date of PD or relapse, occurrence of secondary malignancy, or death from any cause, whichever occurred first. EFS was censored at the date of last disease assessment for patients who were not reported with PD, relapse, occurrence of secondary malignancy or death.
Time Frame: Up to 849 days.
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 2 | 2 | 0 | 2 | 1 | 0
Months | NA [NA to NA] — Median EFS not estimated due to small number of patients per treatment arm. | NA [NA to NA] — Median EFS not estimated due to small number of patients per treatment arm. |  | NA [NA to NA] — Median EFS not estimated due to small number of patients per treatment arm. | NA [NA to NA] — Median EFS not estimated due to small number of patients per treatment arm. |

8. Secondary Outcome: Overall Survival (OS) [in Leukaemia Patients]
Description: Overall survival was defined as time from first infusion of Volasertib to death from any cause. For patients who were lost to follow-up, OS were censored on the last date the patients were known to be alive.
Time Frame: Up to 849 days.
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 2 | 2 | 0 | 2 | 1 | 0
Months | NA [NA to NA] — Median OS not estimated due to small number of patients per treatment arm. | NA [NA to NA] — Median OS not estimated due to small number of patients per treatment arm. |  | NA [NA to NA] — Median OS not estimated due to small number of patients per treatment arm. | NA [NA to NA] — Median OS not estimated due to small number of patients per treatment arm. |

9. Secondary Outcome: Maximum Measured Concentration (Cmax, Norm) of Volasertib
Description: This outcome measure presents dose normalized maximum measured concentration of Volasertib in plasma (Cmax, norm).
Time Frame: Cycle 1: -0:05 (hour/s: minute/s) before drug administration and 1:00, 1:30, 3:00, 24:00, 96:00, 216:00 after drug administration. Cycle >=2: -0:05 (hour/s: minute/s) before drug administration and 1:00 after drug administration.
Population: Pharmacokinetic Set (PKS): All evaluable patients were included in the PK analysis. A patient was considered to be not evaluable, if the patient had an important protocol violation relevant to the evaluation of PK or had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 4 | 0
ng/mL/mg | 5.34 (22.0) | 9.71 (128) | 3.60 (35.1) | 2.46 (54.9) | 2.50 (94.6) |

10. Secondary Outcome: Trough Concentration (Cpre, 2) of Volasertib
Description: This outcome measure presents pre-dose concentration of Volasertib in plasma immediately before administration of the second dose (Cpre,2).
  The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Time Frame: as for outcome 9
Population: Pharmacokinetic Set: All evaluable patients were included in the PK analysis. A patient was considered to be not evaluable, if the patient had an important protocol violation relevant to the evaluation of PK or had insufficient data. The number of participants analysed are the number of participants with available data at the timepoint of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 3 | 2 | 0 | 0 | 0 | 0
ng/mL | 1.48 (60.3) | 1.13 (17.6) |  |  |  |

11. Secondary Outcome: Area Under the Concentration-Time Curve (AUC0-∞, Norm) of Volasertib in Plasma
Description: This outcome measure presents dose normalized area under the concentration-time curve of Volasertib in plasma over the time interval from zero extrapolated to infinity.
Time Frame: as for outcome 9
Population: Pharmacokinetic Set: All evaluable patients were included in the PK analysis. A patient was considered to be not evaluable, if the patient had an important protocol violation relevant to the evaluation of PK or had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 4 | 0
ng*h/mL/mg | 41.7 (40.1) | 51.2 (69.8) | 36.4 (28.2) | 28.6 (19.0) | 22.1 (37.9) |

12. Secondary Outcome: Half-Life (t1/2) of Volasertib
Description: This outcome measure presents half-life of Volasertib.
Time Frame: as for outcome 9
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib 300 mg/m2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 4 | 0
h | 102 (28.6) | 130 (14.1) | 54.8 (27.2) | 78.6 (27.3) | 52.7 (17.7) |

ADVERSE EVENTS:
Time Frame: From the first drug administration until 30 days after the last drug administration.
Description: Treated Set
Groups:
- 2 to <12 Years: Volasertib Pooled Total: The pooled total of patients administered Volasertib 200 mg/m2/250 mg/m2/300 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour on Day 1 of 14-day cycle.
- 12 to <18 Years: Volasertib 250 mg/m2: The patients were administered Volasertib 250 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour on Day 1 of 1-day cycle.
- 12 to <18 Years: Volasertib Pooled Total: The pooled total of patients administered Volasertib 200 mg/m2/250 mg/m2 (solution for infusion) by intravenous infusion over approximately 1 hour on Day 1 of 14-day cycle.
Arm/Group | 2 to <12 Years: Volasertib 200 mg/m2 | 2 to <12 Years: Volasertib 250 mg/m2 | 2 to <12 Years: Volasertib 300 mg/m2 | 2 to <12 Years: Volasertib Pooled Total | 12 to <18 Years: Volasertib 200 mg/m2 | 12 to <18 Years: Volasertib 250 mg/m2 | 12 to <18 Years: Volasertib Pooled Total
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 5/6 | 7/12 | 6/6 | 4/4 | 10/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 12/12 | 6/6 | 3/4 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 to <12 Years: Volasertib 200 mg/m2 (N=3) | 2 to <12 Years: Volasertib 250 mg/m2 (N=3) | 2 to <12 Years: Volasertib 300 mg/m2 (N=6) | 2 to <12 Years: Volasertib Pooled Total (N=12) | 12 to <18 Years: Volasertib 200 mg/m2 (N=6) | 12 to <18 Years: Volasertib 250 mg/m2 (N=4) | 12 to <18 Years: Volasertib Pooled Total (N=10)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 5 | 2 | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bone marrow toxicity (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 to <12 Years: Volasertib 200 mg/m2 (N=3) | 2 to <12 Years: Volasertib 250 mg/m2 (N=3) | 2 to <12 Years: Volasertib 300 mg/m2 (N=6) | 2 to <12 Years: Volasertib Pooled Total (N=12) | 12 to <18 Years: Volasertib 200 mg/m2 (N=6) | 12 to <18 Years: Volasertib 250 mg/m2 (N=4) | 12 to <18 Years: Volasertib Pooled Total (N=10)
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Alanine aminotransferase decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 0 | 2
Antithrombin III decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 2 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Blood pressure increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 2 | 1 | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | 1 | 1 | 2
Platelet count decreased (Investigations) | 1 | 0 | 1 | 2 | 1 | 1 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 2 | 1 | 1 | 2
International normalised ration increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 6 | 2 | 1 | 3
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Cranial nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 2 | 1 | 2 | 3
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
IIIrd nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 2 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 4 | 3 | 1 | 4
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 2
Pyrexia (General disorders) | 2 | 0 | 0 | 2 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 3 | 3 | 1 | 4
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 2 | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.